CLINICAL TRIAL: NCT07127666
Title: Centering Children and Care Partners in Complex Pediatric Hospital Stays: Evaluation of a Structured Inpatient Agenda-setting Intervention for Multidisciplinary Family Meetings
Brief Title: ASKids! Inpatient Agenda-Setting Study for Hospitalized Children With Medical Complexity
Acronym: ASKids
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Catherine Hylas Saunders, Principal Investigator of the Healthcare Experience Lab (HEx Lab), Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY02002855; UM1TR004772 (NIH)
Record Dates: First submitted 2025-08-05; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Medical Complexity
Keywords: clinical agenda-setting; pediatric inpatient care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Implements Structured Agenda-Setting Intervention) (Experimental): The study team will implement a structured clinical visit agenda-setting (SAS) intervention customized for the pediatric inpatient environment.
  Interventions: Other: Structured Agenda-Setting Tool

INTERVENTIONS:
Other: Structured Agenda-Setting Tool — We are testing a novel clinical visit agenda-setting intervention developed through participatory research methods for the pediatric inpatient environment. This structured agenda-setting (SAS) intervention will be co-designed to include structured discussion topic areas with the option for patients (when appropriate) and their care partners to consider and indicate their priority topic areas and take notes before, during, and after a clinical visit.

SUMMARY:
The goal of this open pilot is to co-design and test a clinical agenda-setting intervention in the inpatient pediatric environment. We pilot a co-designed structured agenda-setting intervention (SAS) for multi-family meetings about children with medical complexity. Our open pilot will evaluate the feasibility and acceptability of using the SAS during routine multidisciplinary family meetings (MFM) at Dartmouth Hitchcock Medical Center. By doing an open pilot, researchers will learn if the agenda-setting instrument and implementation process are feasible and acceptable to patients, their care partner and their clinicians.

DETAILED DESCRIPTION:
In this open pilot, the researchers will adapt and administer a novel structured agenda-setting tool (SAS) in the inpatient pediatric environment. The researchers will determine if their procedures for screening eligible participants, administering the intervention, and administering outcome and other questionnaires are appropriate. Learnings from the open pilot will feed forward into procedures in applications for larger trials of the intervention.

This study only has one arm, the intervention arm. The intervention, the co-adapted SAS, will be administered to all enrolled participants.

Future Directions: This open pilot will provide preliminary data for potential future larger trials.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric Inpatients: Children aged 7-17 years
* Can communicate in English
* Able to provide verbal assent, with consent from their care partner
* Dartmouth Hitchcock Medical Center pediatric patient who currently or has recently (within the last 3 months) been hospitalized with a length of stay of 4≥ days Care Partners: - Adults aged 18≥ years
* Can communicate in English
* Able to provide verbal consent
* Care partners of Dartmouth Hitchcock Medical Center pediatric patients who are currently or have recently (within the last 3 months) been hospitalized with a length of stay of 4≥ days

Exclusion Criteria:

* For pediatric inpatients, children < aged 7
* For care partners, children aged <18 years
* Cannot communicate in English
* For pediatric inpatients, unable to provide verbal assent
* For care partners, unable to provide consent
* Prisoners

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Feasibility | Immediately after intervention delivery
  Our primary outcome will be feasibility, assessed by the proportion of patients who receive the intervention.

SECONDARY OUTCOMES:
Primary Process Outcome: Enrollment Rate | Immediately after intervention delivery
  Description: As measured by participant enrollment in REDCap.

OTHER OUTCOMES:
Primary Preliminary Efficacy: Communication Assessment Tool (CAT) | Immediately after intervention delivery
  15-item patient-reported communication tool, with minor context-specific adaptations
Secondary preliminary efficacy: Serious Illness Experience | Immediately after intervention delivery
  Serious illness experience measured by the consideRATE questions; a validated 8-item, plain language (2nd grade) patient-reported experience measure (PREM) with Likert-like response options for patients, and care partners

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth Hitchcock, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
We will de-identified quantitative open pilot data available.
Supporting Information: Study Protocol
Time Frame: The study will use standard processing and documentation protocols adopted by the Inter-university Consortium for Political and Social Research (ICPSR) for data formats, dictionaries, variable names, descriptions, and labels. An XML schema using Data Documenting Initiative standards will also be used for codebooks and other metadata as appropriate. The researchers will share open pilot process and outcomes data in CSV files via openICPSR, which is a self-publishing repository for social, behavioral and health science data and part of the ICPSR.

REFERENCES:
- [Background] Sierpe A, Yen RW, Stevens G, Van Citters AD, Elwyn G, Saunders CH. Agenda-setting in the clinical encounter: A systematic review protocol. PLoS One. 2024 Oct 24;19(10):e0312613. doi: 10.1371/journal.pone.0312613. eCollection 2024. PMID 39446854
- [Background] Saunders CH, Durand MA, Kirkland KB, MacMartin MA, Barnato AE, Elwyn G. Psychometric assessment of the consideRATE questions, a new measure of serious illness experience, with an online simulation study. Patient Educ Couns. 2022 Jul;105(7):2581-2589. doi: 10.1016/j.pec.2022.01.002. Epub 2022 Jan 22. PMID 35260261